CLINICAL TRIAL: NCT05276258
Title: A Randomized Controlled Trial of cryoSPHERE (CRYOS/CRYOS-L) Ablation of Intercostal Nerves for Post-Operative Pain Management in Opioid-Tolerant Patients Undergoing Robotic-Assisted Thoracoscopic Surgery
Brief Title: Cryoablation of Intercostal Nerves for Post-Operative Pain Management in Opioid-Tolerant Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Min P. Kim, MD, Distinguished Professor of Surgery, The Methodist Hospital Research Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO00029370
Record Dates: First submitted 2022-02-14; First posted 2022-03-11 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Pain; Pain, Postoperative
Keywords: pain management; pulmonary surgical procedures; robotic surgical procedures; pneumonectomy; nerve block; neuroma; analgesics, opioid; bupivacaine; length of stay; drug tolerance
MeSH Terms: conditions — Pain; Pain, Postoperative; Agnosia; Neuroma | interventions — Bupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Nerve Block Using Liposomal Bupivacaine and cryoSPHERE Ablation (Experimental): The experimental group (75 participants) will undergo intercostal nerve block using liposomal bupivacaine and the cryoSPHERE ablation of intercostal nerves during robotic-assisted thoracoscopic operation at Houston Methodist Hospital.
  Interventions: Device: cryoSPHERE Ablation; Drug: Bupivacaine
- Historical Controls (Other): A total of 75 propensity score-matched historical controls will be selected from the pool of patients who had standard intercostal nerve block using liposomal bupivacaine alone at Houston Methodist Hospital from January 1, 2017 through January 1, 2022, inclusively.
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Device: cryoSPHERE Ablation — The cryoSPHERE probe will be introduced through a thoracoscopic port and placed inferior to each rib level and 2cm lateral and away from the sympathetic chain when clearly visible or 4cm lateral and away from the spine when the sympathetic chain is not visible. Levels to be ablated are intercostal spaces 3-9. Each intercostal nerve will undergo cryogenic ablation of -70 degrees Celsius for 120 seconds. The probe will be firmly pushed against the nerve for 120 seconds and will only be released from the nerve when the probe has thawed. Axons within the intercostal nerve that send pain signals will be destroyed distal to the cryoablation site. However, the tubules structures (epineurium, perineurium, and endoneurium) of the nerve will remain intact, allowing the axons to regenerate and nerve function to resume after one to three months.
  Other Names: cryoSPHERE
  Arms: Nerve Block Using Liposomal Bupivacaine and cryoSPHERE Ablation
Drug: Bupivacaine — A long needle will be introduced through a thoracoscopic port, and in each intercostal space (1-11), 1ml of liposomal bupivacaine will be injected onto the intercostal nerves to induce intercostal nerve blockage.
  Other Names: liposomal bupivacaine; Exparel

SUMMARY:
The main objective study is to compare the use of the cryoSPHERE probe to the standard-of-care method for pain management of patients receiving robotic-assisted thoracoscopic surgery, including reductions in opioid pain medication use and the development of post-surgical morbidity.

DETAILED DESCRIPTION:
Patients who take more opioid medications after surgery tend to have longer hospital stays, and they are at risk of developing pneumonia and other postoperative morbidities. Opioid-tolerant patients are at a higher risk of developing these morbidities because they often require higher doses of opioid medications to manage their post-operative pain. Reducing post-operative pain in these patients through non-opioid means helps reduce their risk of developing morbidities, and is potentially a more effective form of pain management, particularly in this patient population.

This is a single-center, prospective cohort registry with a historical control, and an estimated duration of 2 years. This study's primary objective is to evaluate the cryoSPHERE probe for ablation in pain control after surgery (measured using opioid medication). The secondary objectives are the evaluation of morbidities, length of stay, cost, and incidence of neuroma formation.

We plan to recruit 75 patients who will receive the cryoSPHERE probe and compare them to 75 patients who did not receive the cryoSPHERE probe. The experimental group will receive cryoSPHERE ablation of intercostal nerves and liposomal bupivacaine. The historical control group will have had robotic-assisted thoracoscopic surgery and an intercostal nerve block with liposomal bupivacaine and no cyroSPHERE probe.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients 18-90 years of age
* Diagnosis requiring robotic-assisted thoracoscopic surgery
* Daily opioid use for at least 30 days consecutively at any point during the last 12 months prior to surgery or using opioids at the time of study enrollment
* Experimental group only: agreement and consent to comply with all aspects of the study protocol and data collection, including follow-up contact.

Exclusion Criteria:

* Previous major surgery at the operative site (thoracotomy)
* Allergy to aluminum
* Allergy to plastics
* Allergy to bupivacaine
* Shingles disease
* Demyelinating illnesses
* Involvement with other interventional studies

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-03-15 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Opioid Use Within 24 Hours After Chest Tube Removal | From the time of chest tube removal to 24 hours after chest tube removal
  Opioid use measured as the daily dose of milligram morphine equivalents (MME)

SECONDARY OUTCOMES:
Total Emergent Adverse Effects (TEAE) | Time of discharge (up to 1 year after surgery), 5 weeks after surgery, 3 months after surgery, and 6 months after surgery
  Morbidity, defined as total emergent adverse effects (TEAE) for the experimental group vs. control
Length of Hospital Stay | From admission to discharge or death, up to 1 year after surgery
  Time spent in the hospital from admission for surgery until discharge or death
Mean Cost of Hospital Care | From admission to discharge or death, up to 1 year after surgery
  Total cost of billed medical care for the surgery
Number of Readmissions | From initial admission for surgery to 28 days after surgery
  The number of readmissions to the hospital
Neuroma Formation | Time of discharge (up to 1 year after surgery), 3 months after surgery, and 6 months after surgery
  The formation of a neuroma around the site of nerve block administration
Pain Score | Time of discharge (up to 1 year after surgery), 5 weeks after surgery, 3 months after surgery, and 6 months after surgery
  Patient's perceived pain level on a scale of 1 to 10
PROMIS3a Pain Intensity | Time of discharge (up to 1 year after surgery), 5 weeks after surgery, 3 months after surgery, and 6 months after surgery
  Patient's perceived pain level on a scale of 3-15, per PROMIS Pain Intensity Short Form 3a v1.0
PROMIS8a Pain Interference | Time of discharge (up to 1 year after surgery), 5 weeks after surgery, 3 months after surgery, and 6 months after surgery
  Patient's perceived pain interference level on a scale of 8-40, per PROMIS Pain Interference Adult Form
Opioid Use after Surgery | Day 1 after surgery, day 3 after surgery, 5 weeks after surgery, 3 months after surgery
  Mean daily opioid use after surgery measured in milligram morphine equivalents (MME)

CONTACTS AND LOCATIONS:
Overall Officials: Min Kim, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Houston Methodist Research Institute, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goto T. What is the best pain control after thoracic surgery? J Thorac Dis. 2018 Mar;10(3):1335-1338. doi: 10.21037/jtd.2018.03.63. No abstract available. PMID 29708130
- [Background] Rice DC, Cata JP, Mena GE, Rodriguez-Restrepo A, Correa AM, Mehran RJ. Posterior Intercostal Nerve Block With Liposomal Bupivacaine: An Alternative to Thoracic Epidural Analgesia. Ann Thorac Surg. 2015 Jun;99(6):1953-60. doi: 10.1016/j.athoracsur.2015.02.074. Epub 2015 Apr 23. PMID 25912739
- [Background] Nobel TB, Adusumilli PS, Molena D. Opioid use and abuse following video-assisted thoracic surgery (VATS) or thoracotomy lung cancer surgery. Transl Lung Cancer Res. 2019 Dec;8(Suppl 4):S373-S377. doi: 10.21037/tlcr.2019.05.14. No abstract available. PMID 32038918
- [Background] Brown LM, Kratz A, Verba S, Tancredi D, Clauw DJ, Palmieri T, Williams D. Pain and Opioid Use After Thoracic Surgery: Where We Are and Where We Need To Go. Ann Thorac Surg. 2020 Jun;109(6):1638-1645. doi: 10.1016/j.athoracsur.2020.01.056. Epub 2020 Mar 3. PMID 32142814
- [Background] Kim MP, Chan EY, Meisenbach LM, Dumitru R, Brown JK, Masud FN. Enhanced recovery after thoracic surgery reduces discharge on highly dependent narcotics. J Thorac Dis. 2018 Feb;10(2):984-990. doi: 10.21037/jtd.2018.01.99. PMID 29607171
- [Background] AtriCure, I., croSPHERE Probe Package Insert.
- [Background] Graves CE, Moyer J, Zobel MJ, Mora R, Smith D, O'Day M, Padilla BE. Intraoperative intercostal nerve cryoablation During the Nuss procedure reduces length of stay and opioid requirement: A randomized clinical trial. J Pediatr Surg. 2019 Nov;54(11):2250-2256. doi: 10.1016/j.jpedsurg.2019.02.057. Epub 2019 Mar 17. PMID 30935731